CLINICAL TRIAL: NCT03243838
Title: Low-dose Apatinib Combined With Neoadjuvant Chemotherapy in the Treatment of Early Triple Negative Breast Cancer (LANCET): A Multicenter, Single-arm, Phase II Trial
Brief Title: Low-dose Apatinib Combined With Neoadjuvant Chemotherapy in the Treatment of Early Triple Negative Breast Cancer
Acronym: LANCET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Kun Wang, Professor, Guangdong Provincial People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20170328
Record Dates: First submitted 2017-08-05; First posted 2017-08-09 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Triple-Negative Breast Cancer
Keywords: Triple-Negative Breast Cancer; apatinib; pCR; OS; Neoadjuvant chemotherapy
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Four cycles of docetaxel combined with apatinib followed by four cycles of epirubicin and cyclophosphamide as Neoadjuvant Treatment for Triple-Negative Breast Cancer
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — All enrolled patients were administered oral apatinib at a dose of 250 mg once daily and intravenously docetaxel (100 mg/m2) every three weeks for four cycles, followed by epirubicin (90 mg/m2) plus cyclophosphamide (600 mg/m2) every three weeks for four cycles. All the treatments were continued until disease progression, patient withdrawal, or unacceptable toxic effects.

SUMMARY:
Triple-negative breast cancer (TNBC) is a special type of breast cancer, endocrine therapy and targeted therapy are completely ineffective, chemotherapy is currently the only effective treatment. How to improve postoperative pathologic complete response（pCR）of neoadjuvant chemotherapy is critical problem to prolong event-free survival (EFS) and overall survival (OS) of TNBC patients. Apatinib is a new oral small molecule tyrosine protease inhibitor, it is effective in inhibiting angiogenesis with a very low concentration. So the standard neoadjuvant chemotherapy regimen of docetaxel and carboplatin combined with apatinib may improve the postoperative pCR and survival outcomes of TNBC patients. Safety and tolerability assessed by number of grade 3 and 4 toxicities and hospitalizations.

DETAILED DESCRIPTION:
All enrolled patients were administered oral apatinib at a dose of 250 mg once daily and intravenously docetaxel (100 mg/m2) every three weeks for four cycles, followed by epirubicin (90 mg/m2) plus cyclophosphamide (600 mg/m2) every three weeks for four cycles. All the treatments were continued until disease progression, patient withdrawal, or unacceptable toxic effects. Granulocyte colony-stimulating factor (G-CSF) used for prophylaxis of febrile neutropenia was permitted according to the American Society of Clinical Oncology (ASCO) guidelines. The biochemical and hematological indexes were evaluated every cycle. Dose modifications of chemotherapy agents, including dose interruptions and dose reductions, were permitted due to certain adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or pathologically confirmed noninflammatory Triple-Negative invasive breast carcinoma (TNBC). The diagnosis of TNBC was defined below: the estrogen receptor and progesterone receptor negativity rates were less than 10%, and the human epidermal growth factor receptor type 2 (HER2) staining was 0 or 1+, and fluorescence in situ hybridization (FISH) detected no HER2 gene amplification
* Clinical stage IIA-IIIB
* Patients must have measurable disease as defined by palpable lesion with caliper and/or a positive mammogram or ultrasound. Bilateral mammogram and clip placement is required for study entry. Baseline measurements of the indicator lesions must be recorded on the Patient Registration Form. To be valid for baseline, the measurements must have been made within the 14 days if palpable. If not palpable, a mammogram or MRI must be done within 14 days. If palpable, a mammogram or MRI must be done within 2 months prior to study entry. If clinically indicated, x-rays and scans must be done within 28 days of study entry.
* Eastern Cooperative Oncology Group(ECOG) performance status 0 to 1 within 14 days of study entry
* Signed informed consent
* Adequate organ function within 2 weeks of study entry: Absolute bone marrow function (hemoglobin concentration of ≥8.0 g/dL, white blood cell count of ≥3000 cells per μL, absolute neutrophil count of ≥1500 cells per μL, platelet count of ≥70000 cells per μL), adequate renal function (creatinine was the upper limit of normal or lower), and adequate liver function (total bilirubin was the upper limit of normal or lower, and aspartate aminotransferase or alanine aminotransferase was twice the upper limit of normal or lower)
* Patients must be aged 18-70 years
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Metastatic disease
* Prior chemotherapy, hormonal therapy, biologic therapy, investigational agent, targeted therapy or radiation therapy for current breast cancer. Patients with history of breast cancer greater than 5 years from initial diagnosis are eligible for the study. Patients may not have received anthracycline-based chemotherapy in the past. Patients with history of ductal carcinoma in situ(DCIS) are eligible if there were treated with surgery alone
* History of previous or current malignancy at other sites with the exception of adequately treated carcinoma in-situ of the cervix or basal or squamous cell carcinoma of the skin. Patients with a history of other malignancies, who remain disease free for greater than five years are eligible
* Uncontrolled blood pressure, previous exposure to apatinib, known allergies to any of the excipients, and a history of unstable angina, myocardial infarction, or class III/IV congestive heart failure (defined by the New York Heart Association) within the past 6 months before day 1 of the trial

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The pathological complete response (pCR) rate in the breast and lymph nodes (ypTis/0ypN0) | up to 24 weeks (at the end of cycle 8, each cycle is 21 days)
  Absence of invasive tumor cells in the breast and lymph nodes and was determined by a local pathologist

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 24 weeks (at the end of cycle 8, each cycle is 21 days)
  ORR was assessed according to RECIST version 1.1, which included patients with measurable disease who achieved a complete or partial response of target lesions.
Event-free survival (EFS) | up to 24 months
  The interval from the start of treatment to progression prior to surgery, post-surgery recurrence, or death due to any cause
Overall survival (OS) | up to 24 months
  The time from registration to death from any cause
Adverse events | up to 24 weeks
  The treatment-related adverse events were assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 (NCI-CTCAE 4.0).

CONTACTS AND LOCATIONS:
Overall Officials: Kun Wang, Study Director — Guangdong Provincial People's Hospital
Locations (2):
- China (2):
  - Guangdong general hospital, Guangzhou, Guangdong
  - Guangdong General Hospital, Guangzhou

REFERENCES:
- [Derived] Yang C, Zhang J, Zhang Y, Ji F, Chen Y, Zhu T, Zhang L, Gao H, Yang M, Li J, Cheng M, Wang K. Low-dose apatinib combined with neoadjuvant chemotherapy in the treatment of early-stage triple-negative breast cancer (LANCET): a single-center, single-arm, phase II trial. Ther Adv Med Oncol. 2022 Aug 12;14:17588359221118053. doi: 10.1177/17588359221118053. eCollection 2022. PMID 35983024